CLINICAL TRIAL: NCT01766466
Title: A Study of the Transition From Cangrelor to Ticagrelor, and Ticagrelor to Cangrelor in Patients With Coronary Artery Disease
Brief Title: Cangrelor Ticagrelor Transition Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: MDCO-CAN-12-03
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — cangrelor; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cangrelor IV + Ticagrelor 180mg at 0.5 hr (Experimental): On Day 1: Open-label cangrelor IV bolus (30 µg/kg), followed by an infusion of 4 µg/kg/min for two hours. Ticagrelor (180 mg) was administered at 0.5 h after the initiation of cangrelor infusion.
  Interventions: Drug: cangrelor; Drug: Ticagrelor
- Cangrelor IV + Ticagrelor 90mg (7 doses) (Experimental): On Day 1: Following completion of cangrelor and ticagrelor dosing, patients were discharged and instructed to take 90 mg ticagrelor every 12 hours for 7 doses (12, 24, 36, 48, 60, 72, and 84 h).
  On Day 5: 12 h post last ticagrelor dose (90 mg), patients received another open-label cangrelor IV bolus (30 µg/kg), followed by an infusion of 4 µg/kg/min for two hours.
  Interventions: Drug: cangrelor; Drug: Ticagrelor
- Cangrelor IV + Ticagrelor 180mg at 1.5 hr (Experimental): On Day 1: Open-label cangrelor IV bolus (30 µg/kg), followed by an infusion of 4 µg/kg/min for two hours. Ticagrelor (180 mg) was administered at 1.5 h after the initiation of cangrelor infusion.
  Interventions: Drug: cangrelor; Drug: Ticagrelor
- Cangrelor IV + Ticagrelor 90mg (6 doses) (Experimental): On Day 1: Following completion of cangrelor and ticagrelor dosing, patients were discharged and instructed to take 90 mg ticagrelor every 12 hours for 6 doses (12, 24, 36, 48, 60, and 72 h).
  On Day 5: 24 h post last ticagrelor dose (90 mg), patients received another open-label cangrelor IV bolus (30 µg/kg), followed by an infusion of 4 µg/kg/min for two hours.
  Interventions: Drug: cangrelor; Drug: Ticagrelor

INTERVENTIONS:
Drug: cangrelor — Open-label cangrelor IV bolus (30 µg/kg), followed by an infusion of 4 µg/kg/min for two hours.
Drug: Ticagrelor — Ticagrelor 180mg dose: administered 0.5 h or 1.5h after the initiation of cangrelor infusion
  Ticagrelor 90mg: 6 or 7 doses (depending on study arm) taken every 12 hours post cangrelor infusion.
  Other Names: Brilinta

SUMMARY:
To demonstrate that patients treated with cangrelor can be directly switched to oral ticagrelor and that patients treated with ticagrelor can be switched to cangrelor without a significant decrease in the extent of inhibition of platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

* greater than / equal to 18 and less than 75 years of age

  1. Previous myocardial infarction defined by admission to the hospital with elevation of markers of injury or the presence of pathologic q waves on at least 2 contiguous electrocardiogram (ECG) leads.

     OR
  2. Previous revascularization by percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery.

     AND
  3. Treatment with aspirin (ASA) 81 mg daily.

     Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Schneider, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The purpose of this study was to study the pharmacodynamic characteristics of transition from IV cangrelor to oral ticagrelor, and ticagrelor to cangrelor in patients with coronary artery disease. This was a single-center study, conducted in Jan-Feb 2013.
Pre-assignment Details: Patients with coronary artery disease who were taking aspirin, but not P2Y12 inhibition were enrolled.
Groups:
- Day 1 - Cangrelor + Ticagrelor (180mg) at 0.5h: Cangrelor IV (2h) + oral ticagrelor (180mg) administered at 0.5h after the initiation of the cangrelor infusion.
- Day 5 - Ticagrelor (90 mg) Dosing (6 Doses): Ticagrelor (90mg) discontinued 24h prior to the initiation of a 2h cangrelor infusion.
- Day 1 - Cangrelor + Ticagrelor (180mg) at 1.5h: Cangrelor IV (2h) + oral ticagrelor (180mg) administered at 1.5h after the initiation of the cangrelor infusion.
- Day 5 - Ticagrelor (90mg) Dosing (7 Doses): Ticagrelor (90mg) discontinued 12h prior to the initiation of a 2h cangrelor infusion.
Period: Day 1
Arm/Group | Day 1 - Cangrelor + Ticagrelor (180mg) at 0.5h | Day 5 - Ticagrelor (90 mg) Dosing (6 Doses) | Day 1 - Cangrelor + Ticagrelor (180mg) at 1.5h | Day 5 - Ticagrelor (90mg) Dosing (7 Doses)
Started | 6 | 0 | 6 | 0
Completed | 6 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Day 5
Arm/Group | Day 1 - Cangrelor + Ticagrelor (180mg) at 0.5h | Day 5 - Ticagrelor (90 mg) Dosing (6 Doses) | Day 1 - Cangrelor + Ticagrelor (180mg) at 1.5h | Day 5 - Ticagrelor (90mg) Dosing (7 Doses)
Started | 0 | 6 | 0 | 6
Completed | 0 | 6 | 0 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ITT Population - Ticagrelor 6 Doses: On Day 1: Open-label cangrelor IV bolus (30 µg/kg), followed by an infusion of 4 µg/kg/min for two hours. Ticagrelor (180 mg) was administered at 0.5 h or 1.5 h after the initiation of cangrelor infusion. Patients were discharged and instructed to take 90 mg ticagrelor every 12 hours for 6 doses.
  On Day 5: Cangrelor was administered after ticagrelor (90 mg)was discontinued 24 hours prior.
- ITT Population - Ticagrelor 7 Doses: On Day 1: Open-label cangrelor IV bolus (30 µg/kg), followed by an infusion of 4 µg/kg/min for two hours. Ticagrelor (180 mg) was administered at 0.5 h or 1.5 h after the initiation of cangrelor infusion. Patients were discharged and instructed to take 90 mg ticagrelor every 12 hours for 7 doses.
  On Day 5: Cangrelor was administered after ticagrelor (90 mg)was discontinued 12 hours prior.
- Total: Total of all reporting groups
Arm/Group | ITT Population - Ticagrelor 6 Doses | ITT Population - Ticagrelor 7 Doses | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.17) | 66.5 (4.32) | 66.4 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Extent of Preservation of Inhibitory Effect Compared With Effect Observed With Cangrelor Alone (at Timepoint 1, Either at 0.5 Hours or 1.25 Hours) or Ticagrelor Alone (Measured 5.25 Hours After Initiation of Cangrelor on Day 1)
Description: A reference point was chosen for comparison and designated the first draw during the cangrelor infusion (0.5 hours or 1.25 hours) as the reference for the effect of cangrelor and designated the final draw on study Day 1 (5.25 hours, or 3.25 hours after cangrelor had been discontinued) as the reference for the effect of ticagrelor. Residual platelet reactivity (the extent of aggregation in the presence or absence of the study drugs) was examined for each of the endpoints using light transmittance aggregometry. Residual platelet reactivity (PR) was measured in response to 20 µmol adenosine diphosphate (ADP) at 300 seconds (final/terminal aggregation response).
Time Frame: Day 1 measures taken at 2 timepoints after cangrelor infusion start: 0.5 or 1.5 hrs (Timepoint 1) and 5.25 hrs (TImepoint 2)
Measure: Mean (Standard Deviation); unit: percentage of platelet reactivity (PR)
Groups:
- Cangrelor + Ticagrelor 180mg at 1.25 h of Cangrelor Infusion; Cangrelor + Ticagrelor 180mg at 0.5 h of Cangrelor Infusion: Cangrelor was administered as IV infusion for 2 hours.
Arm/Group | All Patients | Cangrelor + Ticagrelor 180mg at 1.25 h of Cangrelor Infusion | Cangrelor + Ticagrelor 180mg at 0.5 h of Cangrelor Infusion
Number analyzed (Participants) | 12 | 6 | 6
percentage of platelet reactivity (PR)
  Reference 0.5/1.25 hours - PR | 1.7 (1.7) | 1.3 (2.0) | 2 (1.5)
  1.75 hours - PR | 2.2 (1.4) | 2 (1.8) | 2.3 (1.0)
  2.0 hours - PR | 2.3 (2.2) | 1.2 (1.9) | 3.5 (1.9)

2. Primary Outcome: Extent of Preservation of Inhibitory Effect Compared With Effect Observed During Cangrelor Treatment After Ticagrelor
Description: A reference point was chosen for comparison and designated the first draw during the cangrelor infusion (0.5 hours or 1.25 hours) as the reference for the effect of cangrelor.
  Residual platelet reactivity (the extent of aggregation in the presence or absence of the study drugs) was examined for each of the endpoints using light transmittance aggregometry (LTA). Residual platelet reactivity (PR) was measured in response to 20 µmol ADP at 300 seconds (final/terminal aggregation response).
Time Frame: Day 5 at 1.0 and 2.0 hours after the initiation of cangrelor infusion
Measure: Mean (Standard Deviation); unit: percentage of platelet reactivity (PR)
Arm/Group | All Patients | Ticagrelor Discontinued 24 h Prior to Cangrelor Infusion | Ticagrelor Discontinued 12 h Prior to Cangrelor Infusion
Number analyzed (Participants) | 12 | 6 | 6
percentage of platelet reactivity (PR)
  1.0 hours - PR | 1.5 (1.5) | 1.5 (1.6) | 1.5 (1.5)
  2.0 hours - PR | 1.3 (1.6) | 1.2 (1.5) | 1.5 (1.9)

3. Primary Outcome: Extent of Aggregation Response During Ticagrelor Treatment
Description: Blood samples were taken for platelet function studies to conduct pharmacodynamic assessments including LTA.
  A reference point was chosen for comparison and designated the first draw during the cangrelor infusion (0.5 hours or 1.25 hours) as the reference for the effect of cangrelor and designated the final draw on study Day 1 (5.25 hours, or 3.25 hours after cangrelor had been discontinued) as the reference for the effect of ticagrelor.
  Residual platelet reactivity (PR) (the extent of aggregation in the presence or absence of the study drugs) was examined for each of the endpoints using light transmittance aggregometry. Residual platelet reactivity was measured in response to 20 µmol ADP at 300 seconds (final/terminal aggregation response).
Time Frame: Day 1 at 2.25, 2.5, 2.75, 3 and 4 hrs following initiation of cangrelor infusion
Measure: Mean (Standard Deviation); unit: percentage of platelet reactivity (PR)
Arm/Group | All Patients | Cangrelor + Ticagrelor 180mg at 1.25 h of Cangrelor Infusion | Cangrelor + Ticagrelor 180mg at 0.5 h of Cangrelor Infusion
Number analyzed (Participants) | 12 | 6 | 6
percentage of platelet reactivity (PR)
  Reference 5.25 hours - PR | 4 (3.4) | 2.2 (2.7) | 5.8 (3.1)
  2.25 hours - PR | 12 (11) | 11 (12) | 13 (9.3)
  2.5 hours - PR | 19 (16) | 21 (17) | 16 (15)
  2.75 hours - PR | 10 (9.2) | 7.8 (7.2) | 12 (11)
  3 hours - PR | 7.1 (6.3) | 4.5 (3.4) | 10 (7.6)
  4 hours - PR | 4.6 (3.6) | 2.5 (1.9) | 6.7 (3.7)

ADVERSE EVENTS:
Groups:
- Cangrelor + Ticagrelor 90mg (6 Doses): Ticagrelor was discontinued 24 h prior to cangrelor infusion
- Cangrelor + Ticagrelor 90mg (7 Doses): Ticagrelor discontinued 12 h prior to cangrelor infusion
Arm/Group | Cangrelor + Ticagrelor 90mg (6 Doses) | Cangrelor + Ticagrelor 90mg (7 Doses)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cangrelor + Ticagrelor 90mg (6 Doses) (N=6) | Cangrelor + Ticagrelor 90mg (7 Doses) (N=6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other